CLINICAL TRIAL: NCT05042726
Title: Bilateral Continuous Theta Burst Stimulation of Cerebellum for Drug-refractory Epilepsy: A Double Blind, Randomised, Single Centre, Crossover Clinical Trial
Brief Title: cTBS Targeting Cerebellum for Drug-refractory Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: XijingSN
Record Dates: First submitted 2021-08-31; First posted 2021-09-13 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-08

CONDITIONS: Drug Refractory Epilepsy
Keywords: Drug Refractory Epilepsy; Continuous θ Burst Stimulation; Cerebellar Dentate Nucleus
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS First (Experimental): The first stage, participants received cTBS treatment for a total of 10 times during two weeks, then followed up for eight weeks; the second stage, participants are treated with pseudo-stimulation for a total of 10 times during two weeks, then followed up for 8 weeks similarly.
  Interventions: Device: cTBS First
- Pseudo-stimulation First (Experimental): The first stage, participants received pseudo-stimulation treatment for a total of 10 times during two weeks, then followed up for eight weeks; the second stage, participants are treated with cTBS for a total of 10 times during two weeks, then followed up for 8 weeks similarly.
  Interventions: Device: Pseudo-stimulation First

INTERVENTIONS:
Device: cTBS First — Continuous θ-burst stimulation (cTBS) is characterized by plexus stimulation. The stimulation intensity was 80% resting motor threshold (RMT) at 50Hz of intra plexus pulse while the frequency of inter plexus pulse is 5Hz, the duration was 33.2s, and the number of stimulation pulses was 600. Two groups of stimulation were repeated in each cerebellar dentate nucleus with an interval of 5 min in each group.
  Arms: cTBS First
Device: Pseudo-stimulation First — The transcranial magnetic stimulator operating system has a built-in control group option, in which the stimulation parameters are set consistent with the research group, which can realize the operation of only sound without stimulation.
  Arms: Pseudo-stimulation First

SUMMARY:
This study aims to observe the effect and safety of cerebellar continuous θ burst stimulation (cTBS) for drug-refractory epilepsy(DRE), in order to provide a new treatment for DRE and improve the quality of life of those patients. A total of 44 patients with DRE will have cTBS via accurate navigation to bilateral cerebellar dentate nuclei. Patients will be randomised into 2 groups in a crossover trial design to have 2 week periods of cTBS separated by 8 week washout periods, following which the patient will cross over to have the opposite condition for a further 2 week. Frequency and symptoms of seizures, scalp EEG, clinical scores, and QOLIE-31 were assessed at baseline and after 1 and 2 month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* a) Participants who are in line with the diagnostic criteria for epilepsy,
* b) Participants who are diagnosed as drug-refractory epilepsy,
* c) Participants who has duration of epilepsy ≥2 years and seizure frequency ≥2 times per month,
* d) The type and dosage of anti-epileptic drugs do not change during the experiment,
* e) Participants or their families reject invasive therapy, such as operation,
* f) Participants and their families are aware of this study and sign informed consent.

Exclusion Criteria:

* a) Participants who are in status epilepticus,
* b) Participants who are complicated with serious infection, cerebrovascular disease, malignant tumor and other nervous system diseases, with serious dysfunction of heart, liver, kidney and other organs, and with psychiatric disorders,
* c) Participants who are diagnosed as syncope, hysteria or other non-epileptic attacks,
* d) Participants who are in pregnancy or lactating,
* e) Participants who have incomplete clinical data,
* f) Patients have contraindications of repeated transcranial magnetic stimulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
seizure reduction rate in pre- and post-treatment | 8 weeks
  A 28-day baseline for seizure frequency will be recorded by the patients themselves or their relatives before therapy and then compare to the frequency at 4-week and 8-week after treatment, finally, the rate of reduction in seizure frequency was obtained
responder rate | 8 weeks
  proportion of people with a 50% or greater reduction in seizure frequency following the treatment period

SECONDARY OUTCOMES:
QOLIE-31 scale scores | 8 weeks
  Quality of Life in Epilepsy-31. Scores range from 0 to 100, with higher scores indicating better quality of life.
scalp electroencephalogram | 8 weeks
  Routine scalp electroencephalogram at 40 min
IQ | 8 weeks
  Wechsler Abbreviated Scale of Intelligence. Above 130 points very excellent, 120-129 excellent, 110-119 above average, 90-109 average, 80-89 below average, 70-79 critical level, below 69 mental retardation, 50-69 mild mental retardation, 35-49 moderate mental retardation, 20-34 severe mental retardation, less than 20 extremely severe mental retardation.
MQ | 8 weeks
  Wechsler Memory Scale. Above 130 points very excellent, 120-129 excellent, 110-119 above average, 90-109 average, 80-89 below average, 70-79 critical level, below 69 mental retardation, 50-69 mild mental retardation, 35-49 moderate mental retardation, 20-34 severe mental retardation, less than 20 extremely severe mental retardation.
MoCA | 8 weeks
  Montreal Cognitive Assessment. A max score is 30 points, and a score ≥ 26 is considered normal.
MMSE | 8 weeks
  Mini-Mental State Examination. The normal values are defined as: illiterates >17, primary school >20, junior high school or above >24.
HAMD | 8 weeks
  Hamilton Depression Scale. Total score <7 means normal; between 7 and 17 means possible depression; between 17 and 24 , definitely have depression; >24 means severe depression.
HAMA | 8 weeks
  Hamilton Anxiety Scale. The total score ≥29 may be severe anxiety; ≥21, obvious anxiety; ≥14, definite anxiety; ≥7, may have anxiety; If the score <7, there are no symptoms of anxiety.
SCL-90 | 8 weeks
  Self-reporting Inventory. The total symptom index scores ranged from 1 to 1.5, indicating that the subjects did not feel the symptoms listed in the scale. Between 1.5 and 2.5, indicates that the subject feels a little symptomatic, but not occur frequently. Between 2.5 and 3.5, indicates that the subject feels symptoms, and is mild to moderate. The score between 3.5 and 4.5 indicates that the subjects feel symptoms, and the degree was moderate to severe. A score between 4.5 and 5 indicates that the subject feels symptoms, and the frequency and intensity are very severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Theodore WH, Spencer SS, Wiebe S, Langfitt JT, Ali A, Shafer PO, Berg AT, Vickrey BG. Epilepsy in North America: a report prepared under the auspices of the global campaign against epilepsy, the International Bureau for Epilepsy, the International League Against Epilepsy, and the World Health Organization. Epilepsia. 2006 Oct;47(10):1700-22. doi: 10.1111/j.1528-1167.2006.00633.x. PMID 17054693
- [Background] Forsgren L, Beghi E, Oun A, Sillanpaa M. The epidemiology of epilepsy in Europe - a systematic review. Eur J Neurol. 2005 Apr;12(4):245-53. doi: 10.1111/j.1468-1331.2004.00992.x. PMID 15804240
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] George MS, Aston-Jones G. Noninvasive techniques for probing neurocircuitry and treating illness: vagus nerve stimulation (VNS), transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS). Neuropsychopharmacology. 2010 Jan;35(1):301-16. doi: 10.1038/npp.2009.87. PMID 19693003
- [Background] Hsu WY, Cheng CH, Lin MW, Shih YH, Liao KK, Lin YY. Antiepileptic effects of low frequency repetitive transcranial magnetic stimulation: A meta-analysis. Epilepsy Res. 2011 Oct;96(3):231-40. doi: 10.1016/j.eplepsyres.2011.06.002. Epub 2011 Jun 29. PMID 21715144
- [Background] Cooper YA, Pianka ST, Alotaibi NM, Babayan D, Salavati B, Weil AG, Ibrahim GM, Wang AC, Fallah A. Repetitive transcranial magnetic stimulation for the treatment of drug-resistant epilepsy: A systematic review and individual participant data meta-analysis of real-world evidence. Epilepsia Open. 2017 Dec 27;3(1):55-65. doi: 10.1002/epi4.12092. eCollection 2018 Mar. PMID 29588988
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Koc G, Gokcil Z, Bek S, Kasikci T, Eroglu E, Odabasi Z. Effects of continuous theta burst transcranial magnetic stimulation on cortical excitability in patients with idiopathic generalized epilepsy. Epilepsy Behav. 2017 Dec;77:26-29. doi: 10.1016/j.yebeh.2017.09.011. Epub 2017 Oct 23. PMID 29073474
- [Background] Brighina F, Daniele O, Piazza A, Giglia G, Fierro B. Hemispheric cerebellar rTMS to treat drug-resistant epilepsy: case reports. Neurosci Lett. 2006 Apr 24;397(3):229-33. doi: 10.1016/j.neulet.2005.12.050. Epub 2006 Jan 19. PMID 16426754
- [Background] Krook-Magnuson E, Szabo GG, Armstrong C, Oijala M, Soltesz I. Cerebellar Directed Optogenetic Intervention Inhibits Spontaneous Hippocampal Seizures in a Mouse Model of Temporal Lobe Epilepsy. eNeuro. 2014 Dec;1(1):ENEURO.0005-14.2014. doi: 10.1523/ENEURO.0005-14.2014. PMID 25599088